CLINICAL TRIAL: NCT00992875
Title: Does Mindfulness Training Change the Processing of Social Threat?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mind and Life Institute, Hadley, Massachusetts (Other); European Commission (Other)
Responsible Party: Principal Investigator, Britta Holzel, Research Fellow, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2008A057212; FP7-PEOPLE-IOF-2008: 236975
Record Dates: First submitted 2009-09-28; First posted 2009-10-09 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Healthy; Stress
Keywords: Healthy but stressed individuals
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — Behavioral intervention, mindfulness meditation in form of yoga, sitting meditation, body scan and mindfulness to routine activities

SUMMARY:
Training in mindfulness, the non-judgmental observation of experiences as they arise in the present moment, has been increasingly and successfully applied to the treatment of normative stress conditions and mental disorders. Yet, the neurological mechanisms that underlie the reported improvements are still largely unknown. This longitudinal study will investigate the influence of mindfulness training on a key underpinning of mental health, namely emotion regulation, and its associated brain activity. Healthy participants will be randomly assigned to either a validated eight week Mindfulness-based stress reduction (MBSR) program or to a control condition. In a pre-post investigation, participants' subjective reactions to aversive emotional stimuli (affective facial expressions) will be assessed, as will the associated brain activation using functional magnetic resonance imaging (fMRI). The investigators hypothesize that after the training the MBSR participants will rate the pictures as less aversive compared to control participants. Furthermore, the MBSR participants will show a patter of brain activation indicative of improved emotion regulation, relative to control participants. Finally, the effect of MBSR on the gray matter structure of the brain will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* no previous significant meditation or yoga experience
* eligible for MRI scanning (no metallic implants, not pregnant, not claustrophobic)
* no significant previous meditation or yoga experience

Exclusion Criteria:

* DSM-IV diagnosis for depression, manic episodes, GAD, social phobia, anorexia, bulimia, schizophrenia, ADHD, substance dependency/abuse, suicidality
* ineligible for MRI scanning (metallic implants, pregnant, claustrophobic)

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
BOLD signal on a 1.5T MRI scanner | the second time-point will take place eight weeks after the first data collection

CONTACTS AND LOCATIONS:
Overall Officials: Sara W Lazar, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

REFERENCES:
- See also: Related Info — http://www.nmr.mgh.harvard.edu/~lazar/Participate.html